CLINICAL TRIAL: NCT00301509
Title: Outcome of Decompensated Hepatitis C Virus-Related Cirrhotic Patients Treated With Peginterferon Alfa-2b and Ribavirin: Results of a Controlled Study
Brief Title: Antiviral Therapy in Decompensated Hepatitis C Virus (HCV) Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 630/DS
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2006-03-13 (Estimated); Status verified 2005-12

CONDITIONS: Liver Cirrhosis, Experimental
MeSH Terms: conditions — Liver Cirrhosis, Experimental | interventions — Ribavirin

INTERVENTIONS:
Drug: peginterferon and ribavirin

SUMMARY:
To evaluate:

1. the impact of combined antiviral therapy (Peginterferon plus ribavirin) on natural history of patients affected with HCV decompensated cirrhosis, after sustained virological response. A controlled study.
2. safety and efficacy of antiviral therapy in this population by using a statistically significally number of patients as controls.

DETAILED DESCRIPTION:
Decompensated HCV cirrhosis is a relevant problem as its clinical evidences predisposes to an high mortality risk, with a survival rate of 50% at 5 years (1,2). Davis et. al processed a mathematical model of the natural history of chronic hepatitis C and projected the total number of cases with cirrhosis increased by more than 50% by 2010 and then plateaued (3). As a result, there will be a dramatic increase in the number of cases with complications of liver failure and decompensated events of cirrhosis will increase to 25% in 2010, 32% in 2020, 36% in 2030, and 38% in 2040 (3, table 1).Liver transplantation is the treatment of choice but the limited number of organ donor makes not realizable for the major of patients. Furthermore, age over 65 years correlated disease is not accepted to enter into the list of liver transplant. To prevent these patients from worsening their liver disease has positive economic implications in terms of health care resources used as diagnostic tests, clinic visits, drug therapy, hospitalization for management of complications, and later on, liver transplantation, and indirect costs related to lost work time and impaired quality of life. our controlled study on antiviral treatment of decompensated cirrhotics has shown that HCV clearance by therapy can be life-saving, improves hepatic function, and reduces disease progression. Treatment should be encouraged in CTP classes A and B, and especially in patients infected by genotype 2. The benefit of treating patients with genotype 1 remains unproven.

ELIGIBILITY:
Inclusion Criteria: HCV cirrhotics admitted to hospital for a decompensated event, such as ascites, variceal bleeding, and hepatic encephalopathy -

Exclusion Criteria: rapid deterioration of liver and/or renal function, detection of hepatocarcinoma, infection with HIV or HBV viruses, current alcohol or drug abuse, chronic invalidating disease, bacterial infections, platelets <35,000 cells/μL, neutrophils <1,000 cells/μL, haemoglobin level <10 g/dL, total bilirubin >3 mg/dL, and serum creatinine >2.0 mg/dL.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Andriulli, Chief, Principal Investigator — CSS
Locations (1):
- Department of Hepatogastroenterology, CSS, San Giovanni Rotondo, Foggia, Italy